CLINICAL TRIAL: NCT02629120
Title: High Dose Peripheral Blood Stem Cell Transplantation With Post Transplant Cyclophosphamide for Patients With Chronic Granulomatous Disease
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160032; 16-I-0032
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-06-20

CONDITIONS: Chronic Granulomatous Disease Transplant
Keywords: The National Marrow Donor Program (NMDP); Matched Unrelated Donor (MUD); HLA Matched Related Donor
MeSH Terms: interventions — Alemtuzumab; Busulfan; Sirolimus; Cyclophosphamide; Whole-Body Irradiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Active Comparator): There is only one treatment arm for this study
  Interventions: Drug: Alemtuzumab; Drug: Busulfan; Drug: Sirolimus; Drug: Cyclophosphamide; Radiation: Total Body Irradiation; Biological: Peripheral blood stem cells

INTERVENTIONS:
Drug: Alemtuzumab — Transplant Conditioning Drug: Monoclonal antibody that targets recipient and donor T-cells to prevent graft verses host disease. Not an IND. This is a well studied drug, and is not under an IND.
Drug: Busulfan — Transplant Conditioning Drug: Chemotherapy to create space in the patient's bone marrow so that the donor peripheral blood stem cells can repopulate in the patient's bone marrow. This is a well studied drug, and is not under an IND.
Drug: Sirolimus — Immunosuppressant to prevent donor peripheral blood stem cell rejection and graft versus host disease. This is a well studied drug, and is not under an IND.
Drug: Cyclophosphamide — Post transplant cyclophosphamide given to prevent graft verses host disease. This is a well studied drug, and is not under an IND.
Radiation: Total Body Irradiation — Transplant Conditioning Total Body Radiation (300cGy in 2 fractionated doses), given only to patient receiving matched unrelated donor cells, to create space in the patient's bone marrow so that the donor peripheral blood stem cells can repopulate in the patient's bone marrow.
Biological: Peripheral blood stem cells — Donor Peripheral blood stem cells, either matched unrelated donor or matched related relative to replace the patient's immune cells with functional immune cells. The peripheral blood stem cells are not regulated by the FDA.

SUMMARY:
Chronic granulomatous disease (CGD) affects white blood cell function. Currently, the only curative treatment is bone marrow transplant to replace the abnormal stem cells with new ones (donor cells) capable of making a normal immune system. Transplant problems include graft versus host disease (GvHD) and graft rejection. With GvHD, donor cells attack the recipient s normal tissue. Researchers want to use preparation drugs and a high cell dose to increase graft success. They want to use 2 immunosuppressive drugs (cyclophosphamide and sirolimus) to lessen the risk of GvHD.

DETAILED DESCRIPTION:
Study Description:

Alemtuzumab, targeted busulfan, and TBI, with a 10/10 related or MUD donor graft or a 9/10 single HLA mismatch graft followed by post-transplant cyclophosphamide.

Primary Objectives:

To determine engraftment rates with the use of high cell doses, without increasing the risk of GvHD by using post-transplant cyclophosphamide and sirolimus in conjunction with a busulfan based conditioning regimen. We will compare the incidence of graft rejection/failure and GvHD to the incidence obtained from Protocol 07-I-0075.

Secondary Objectives:

To measure the engraftment rate and the engraftment kinetics using such a regimen.

To assess the level and kinetics of immune reconstitution (via chimerism) when using post- transplant cyclophosphamide.

To further elucidate the factors involved in the development of GvHD and graft rejection/failure.

To evaluate the risk of viral infections in the setting of Alemtuzumab (Campath-1H) and post-transplant cyclophosphamide.

Primary Endpoint:

Reduced incidence of graft failure or rejection (as defined by >20% engraftment by oxidase- positive neutrophils in at least 95% of participants by Day 100, 6 months, and 1 year post BMT) will be assessed as event-free survival (EFS). Graft failure will result in disease recurrence. This will be assessed in a composite form along with GvHD (see Biostatistical Considerations section 17).

Secondary Endpoints:

Same or reduced rate of grade 3-4 aGvHD of <20% .

Establish stable mixed chimerism.

Improve rapidity of immune reconstitution.

Overall survival.

Tertiary Endpoints:

Evaluation of inflammatory markers as risk factors for

engraftment syndrome

ELIGIBILITY:
* INCLUSION CRITERIA:
* Must have confirmed Chronic Granulomatous Disease.
* Must have sufficient complications from underlying disease to warrant undergoing transplantation (either a history of or ongoing inflammation/CGD related autoimmunity OR a CGD related infection while on prophylaxis) OR or have a Quartile 1 and/or 2 residual oxidase production level.
* Ages 4 years - 65 years
* HLA-matched family donor graft or an HLA matched unrelated peripheral blood stem cell (PBSC) graft (10/10 or 9/10 mismatch) available
* Must be HIV negative
* When discharged from the hospital must be able to stay within one hour s travel of the NIH for the first 3 months after transplantation and have a family member or other designated companion to stay with during the post transplant period.
* Must provide a durable power of attorney for health care decisions to an appropriate adult relative or guardian in accordance to NIH -200 NIH Durable Power of Attorney for Health Care Decision Making .
* If of child-bearing potential, must agree to consistently use contraception from one month prior to, and throughout, study participation, and for 3 months post-study. Acceptable forms of contraception are:

  * Contraceptive pills or patch, Norplant , Depo-Provera , or other FDA-approved contraceptive method
  * Male partner has previously undergone a vasectomy.
  * Male participants will be advised to consistently use contraception throughout study participation and for 3 months post-transplant.

EXCLUSION CRITERIA:

* Eastern Cooperative Oncology Group (ECOG) or equivalent performance status greater than or equal to 3 (See Supportive Care guidelines, available at http://intranet.cc.nih.gov/bmt/clinicalcare)
* Left ventricular ejection fraction < 40%
* Transaminases > 5x upper limit of normal based on the participant s clinical situation and at the discretion of the investigator
* Psychiatric disorder or mental deficiency severe enough as to make compliance with the HSCT treatment unlikely, and/or making regulatorily and legally effective informed consent impossible
* Major anticipated illness or organ failure incompatible with survival from AlloPBSC transplant
* Pregnant or lactating
* HIV positive
* Uncontrolled seizure disorder
* Individuals older than 65 are excluded. It is known from standard transplantation that these participants have a higher risk of morbidity and mortality related to transplantation. Given the investigational nature of this protocol, the risk benefit ratio is not warranted to include these participants at this time.
* Any condition or circumstance which the PI feels would create difficulty in maintaining compliance with the requirements of this protocol.
* Individuals who are not willing to submit their information as part of the Alemtuzumab (Campath) Distribution Program application or participants whom the Distribution Program committee has determined are not qualified to receive alemtuzumab.

  --NOTE: Alemtuzumab (Campath-1H) (intravenous [IV] formulation) is no longer distributed commercially. In order to receive product, the physician must contact the program for the patient. If the patient is not willing to consent to submit their info (demographics, contact information, and rationale for use) to the program such that we can obtain the drug, then we cannot proceed with conditioning; therefore no transplant will occur on this protocol.
* Patients with a CRP greater than 100 mg/L within 30 days of anticipated transplant.

  * If the underlying inflammation is controlled for one month with repeat CRP testing showing a level of less than 100 on at least two separate testings, the patient will be reconsidered for transplant. If during this time period a CRP of greater than 100 is measured, then the patient would no longer be eligible for transplant.

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
To determine engraftment rates with the use of high cell doses, without increasing the risk of GvHD by using post-transplant cyclophosphamide and sirolimus in conjunction with a busulfan- based conditioning regimen. We will compare the incidence... | 5 years
  This study is still recruiting patients.

SECONDARY OUTCOMES:
To measure the engraftment rate and the engraftment kinetics using such a regimen | 5 years
  This study is still recruiting patients
To assess the level and kinetics of immune reconstitution (via chimerism) when using post- transplant cyclophosphamide | 5 years
  This study is still recruiting patients
To further elucidate the factors involved in the development of GvHD and graft rejection/failure | 5 years
  This study is still recruiting patients

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Kang, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The following data will be shared: @@@@@@@@@@@@All the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data availability and the duration of the data availability are as follows:@@@@@@@@@@@@Transplant data shared with CIBMTR, BTRIS, and the NML will be shared at the onset of signing the protocol and will be maintained in shared databases with no end date. @@@@@@@@@@@@Transplant data submitted for publication will be immediately available following publication with no end date.
Access Criteria: IIndividual deidentified data will be shared with: @@@The Center for International Blood and Transplant Research (CIBMTR), as required by the Stem Cell Therapeutic and Research Act of 2005 https://www.congress.gov/bill/109th-congress/house-bill/2520 @@@An NIH-funded or approved public repository. @@@Publications@@@Public presentations. @@@Individual identified participant data will be shared with: @@@Approved outside collaborators under appropriate agreements, such as the Neutrophil Monitoring Lab (NML) in Frederick, Md.@@@Biomedical Translational Research Information System (BTRIS).@@@The following related documents will be available:@@@Study Protocol @@@Statistical analysis plan @@@Analytic code@@@CIBMTR, BTRIS, and the NML data will be shared at the onset of signing the protocol and will be maintained in shared databases with no end date. @@@Data submitted for publication will be immediately available following publication with no end date.@@@

REFERENCES:
- [Background] Kottaridis PD, Milligan DW, Chopra R, Chakraverty RK, Chakrabarti S, Robinson S, Peggs K, Verfuerth S, Pettengell R, Marsh JC, Schey S, Mahendra P, Morgan GJ, Hale G, Waldmann H, de Elvira MC, Williams CD, Devereux S, Linch DC, Goldstone AH, Mackinnon S. In vivo CAMPATH-1H prevents graft-versus-host disease following nonmyeloablative stem cell transplantation. Blood. 2000 Oct 1;96(7):2419-25. PMID 11001893
- [Background] Kang EM, Hsieh MM, Metzger M, Krouse A, Donahue RE, Sadelain M, Tisdale JF. Busulfan pharmacokinetics, toxicity, and low-dose conditioning for autologous transplantation of genetically modified hematopoietic stem cells in the rhesus macaque model. Exp Hematol. 2006 Feb;34(2):132-9. doi: 10.1016/j.exphem.2005.10.010. PMID 16459181
- [Background] Horwitz ME, Barrett AJ, Brown MR, Carter CS, Childs R, Gallin JI, Holland SM, Linton GF, Miller JA, Leitman SF, Read EJ, Malech HL. Treatment of chronic granulomatous disease with nonmyeloablative conditioning and a T-cell-depleted hematopoietic allograft. N Engl J Med. 2001 Mar 22;344(12):881-8. doi: 10.1056/NEJM200103223441203. PMID 11259721
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-I-0032.html